CLINICAL TRIAL: NCT02144532
Title: Effectiveness of Wearing a Compression Garment (SED CICATREX® Model) for Patients With Hypermobility Type of Ehlers-Danlos Syndrome
Brief Title: Wearing a Compression Garment for Patients With Hypermobility Type of Ehlers-Danlos Syndrome
Acronym: VETCOSED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-755
Record Dates: First submitted 2014-05-07; First posted 2014-05-22 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Ehlers-Danlos Syndrome Hypermobility Type
Keywords: Ehlers-Danlos syndrome; hypermobility; Compression garment; pain; isokinetic evaluation
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3; Ehlers-Danlos Syndrome; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with EDS hypermobility type (Experimental): Patients with EDS hypermobility type wearing compression garment then compression garment removal
  Interventions: Device: short-sleeved vest CICATREX SED®)

INTERVENTIONS:
Device: short-sleeved vest CICATREX SED®) — Each patient wears a compression custom-made garment (short-sleeved vest CICATREX SED®) according to the medical prescription during the first 4 weeks (BEFORE phase). Then each patient should not wear the compression garment for the next 4 weeks (AFTER phase).

SUMMARY:
The Ehlers-Danlos syndrome (EDS) is a rare genetic disease caused by an anomaly of the connective tissue. This syndrome has different forms. Hypermobility type is the most common. It is characterized by generalized joint hypermobility, associated with a chronic pain syndrome. Pains appear as the most frequent demonstration of this syndrome, the worst lived and the most crippling.

Faced with insufficient effect of drug treatment, other alternatives have been proposed to relieve these patients. Compression garments have been developed. They appear as medical devices targeted specifically for patients with hypermobility EDS type: in the symptomatic treatment of joint pain, in stabilizing joints by proprioceptive effect and of muscle globulization, and in the functional improvement.

The VETCOSED study is a quasi-experimental study of type "Before / After", monocentric, open. The study is realized in the Centre Médico-Chirurgical et de Réadaptation des Massues - Croix Rouge Française de Lyon, in association with the Pôle Information Médicale Evaluation Recherche des Hospices Civils de Lyon. This study concerns about 40 patients with EDS hypermobility type, which will be followed for 8 weeks: 4 weeks during which they will wear a compression custom-made garment (short-sleeved vest CICATREX SED®), and 4 weeks during which they do not carry this garment.

The main objective is to demonstrate the effectiveness of compression garments in the EDS hypermobility type, especially in terms of symptomatic improvement joint pain.

The main outcomes expected of this study are:

* an improvement of the power and the peaks of couple of muscles rotators of shoulders.
* a decrease of the pains and the defects of articular stability of the shoulder
* an improvement of the quality of life and the functional independence of these patients

ELIGIBILITY:
Inclusion Criteria:

* Ehlers-Danlos syndrome hypermobility type confirmed the diagnosis of a geneticist
* with an instability of one or both shoulders, painful or considered invalidating by the patient (recurrent dislocation or subluxation : at least once / month or at least 12 times / year)
* having a joint hypermobility syndrome (abnormal mobility and in a non-physiological axis), with a Beighton score of greater than or equal to 5 of 9
* age greater than or equal to 18 years
* size greater than or equal to 1 m 40
* sufficient understanding of the French language in order to respond to self-report questionnaires

Exclusion Criteria:

* hyperalgic episode in progress
* unstable cardiac disease
* previous history of shoulder surgery
* severe skin lesions,
* pregnancy in progress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Power (in watts) of the external rotators of the shoulder of the dominant arm measured by concentric isokinetic evaluation at a constant angular velocity of 180 °/s | 2 months follow-up
  The evaluations will be conducted 3 times:
  * at the inclusion (D0)
  * at the end of the BEFORE phase (4 weeks with the compression garment: D0 + 28)
  * at the end of the AFTER phase (4 weeks without the compression garment: D0 + 56) For each measurement, evaluations will be made with then without the compression garment.

SECONDARY OUTCOMES:
Level of pain expressed in the shoulders of patients | D0,D28,D56
  Evaluation of the level of pain each month by the physician investigator on Visual Analogue Scale :
  * at the inclusion (D0)
  * at the end of the BEFORE phase (4 weeks with the compression garment: D0 + 28)
  * at the end of the AFTER phase (4 weeks without the compression garment: D0 + 56)
Score of quality of life measured by the medical outcomes study Short-Form General Health Survey (SF-36 scale) | D0,D28,D56
  The score of quality of life is measured by self-administered questionnaire (SF-36 scale) at each follow-up visit:
  * at the inclusion (D0)
  * at the end of the BEFORE phase (4 weeks with the compression garment: D0 + 28)
  * at the end of the AFTER phase (4 weeks without the compression garment: D0 + 56)
Score of satisfaction measured by the Quebec User Evaluation of Satisfaction with assistive Technology (QUEST) | D0,D28,D56
  The score of satisfaction is measured by self-administered questionnaire (QUEST) at each follow-up visit:
  * at the inclusion (D0)
  * at the end of the BEFORE phase (4 weeks with the compression garment: D0 + 28)
  * at the end of the AFTER phase (4 weeks without the compression garment: D0 + 56)
Functional independence score measured by Health Assessment Questionnaire (HAQ) | D0,D28,D56
  The score of functional independence is measured by self-administered questionnaire (HAQ) at each follow-up visit:
  * at the inclusion (D0)
  * at the end of the BEFORE phase (4 weeks with the compression garment: D0 + 28)
  * at the end of the AFTER phase (4 weeks without the compression garment: D0 + 56)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle CHALEAT-VALAYER, MD, Principal Investigator — Médecine Physique et de Réadaptation, Centre Médico-Chirurgical de Réadaptation des Massues
Locations (1):
- Médecine Physique et de Réadaptation, Centre Médico-Chirurgical de Réadaptation des Massues - Croix-Rouge française, Lyon, France